CLINICAL TRIAL: NCT03672097
Title: Phase IV, Non-comparative, Open Label, Multicenter, 28-Week Switching Study of Prasugrel Maintenance Dose From Clopidogrel in Patients With Acute Coronary Syndrome (ACS) Who Underwent a Percutaneous Coronary Intervention (PCI) in Taiwan
Brief Title: Prasugrel Switching Study in Patients With Acute Coronary Syndrome (ACS) Who Underwent Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo Taiwan Ltd., a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS747S-B-A4003
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Results first posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-10

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Percutaneous Coronary Intervention (PCI); ST elevation myocardial infarction (STEMI); Non-ST elevation myocardial infarction [NSTEMI]; Unstable angina (UA); Prasugrel; ACS-PCI
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Angina, Unstable | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prasugrel (Experimental): Participants with ACS who underwent PCI, and were previously taking clopidogrel, receive a maintenance dose (MD) of prasugrel for a total of 28 weeks (optionally up to a maximum 12 months of P2Y12 inhibitor treatment after ACS underwent PCI)
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Prasugrel — Prasugrel, oral tablets, containing 3.75 mg per tablet
  Other Names: Efient®

SUMMARY:
This Phase IV, multicenter trial is designed to assess the efficacy of prasugrel in preventing the formation of blood clots in Taiwanese patients with ACS who have been treated with PCI.

ELIGIBILITY:
Inclusion Criteria:

* Is within the age limits and has signed informed consent
* Weighs at least 50 kg
* Had a previous diagnosis of ACS (UA, STEMI, or NSTEMI), underwent PCI, and received one of the following treatments:

  * Clopidogrel MD of 75 mg and aspirin 81-100 mg for 2-8 weeks following clopidogrel loading dose (LD) of 300 mg or 600 mg at the time of PCI
  * Ticagrelor MD of 90 mg twice daily (BID) and aspirin 81-100 mg for 1-4 weeks and switching to clopidogrel MD of 75 mg and aspirin 81-100 mg for 2-4 weeks following ticagrelor LD of 180 mg at the time of PCI
  * Clopidogrel MD 75 mg and aspirin 81-100 mg for 2-8 weeks following ticagrelor LD of 180 mg at the time of PCI
  * Or based on investigator's judgment with at least 2 weeks continued use of clopidogrel MD and aspirin 81-100 mg per day before switching to prasugrel and maximum 8 weeks P2Y12 inhibitors MD treatment (prasugrel is not allowed)
* Is willing and able to abide by the rules of the research unit and study restrictions
* If a woman of child-bearing potential, has a negative serum pregnancy test at screening
* Agrees to use at least one method of contraception during the study

Exclusion Criteria:

* Has active bleeding, significant risk of hemorrhage, or unusual susceptibility to bleed
* Had previous hemorrhagic stroke at any time, or transient ischemic attack (TIA) or ischemic stroke within 3 months before the informed consent date
* Has known allergies or hypersensitivity to prasugrel, aspirin, or any of their excipients
* Has significant hypertension at screening or baseline assessment
* Has hemoglobin levels <10.5 g/dL or hematocrit levels <30%
* Has severe left ventricular systolic dysfunction, ejection fraction <30%
* Is currently undergoing hemodialysis
* Has evidence of severe hepatic disease or any of the following: serum alanine transaminase or aspartate transaminase ≥3 times the upper limit of normal (ULN); or bilirubin ≥2 times the ULN at screening
* Has any clinical laboratory result performed at screening that is determined to be detrimental to the patient or could compromise the study as determined the Investigator
* Has previously participated in this study or in another interventional trial that is not compatible with this study
* Has evidence of significant active neuropsychiatric disease, alcohol abuse or drug abuse as determined by the Investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (10):
- Taiwan (10):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Cheng Hsin General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Liu PY, Su CH, Kuo FY, Lee WL, Wang YC, Lin WS, Chu PH, Lu TM, Lo PH, Lee CH, Lan WR, Huang CL, Tsukiyama S, Yang WC, Cheng LC, Rafael V, Nikolajsen C, Yin WH. Prasugrel switching from clopidogrel after percutaneous coronary intervention for acute coronary syndrome in Taiwanese patients: an analysis of safety and efficacy. Cardiovasc Interv Ther. 2022 Apr;37(2):269-278. doi: 10.1007/s12928-021-00771-w. Epub 2021 Apr 4. PMID 33813727

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 204 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 10 clinic sites in Taiwan from 01 Nov 2018 to 19 Aug 2020. One patient did not receive study treatment.
Pre-assignment Details: Participants with a previous diagnosis of acute coronary syndrome (ACS) who had undergone percutaneous coronary intervention (PCI) and had been previously treated with a maintenance dose of clopidogrel.
Groups:
- Prasugrel: Participants with ACS who underwent PCI, and were previously taking clopidogrel, who received a maintenance dose of prasugrel for a total of 28 weeks (optionally up to a maximum 12 months of P2Y12 inhibitor treatment after ACS participants underwent PCI).
Period: Period 1
Arm/Group | Prasugrel
Started | 204
Completed | 200
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Did not receive treatment | 1
Period: Period 2
Arm/Group | Prasugrel
Started | 200
Completed | 196
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: The baseline demographics were reported from the Safety Population.
Arm/Group | Prasugrel
Number analyzed (Participants) | 203
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 130
  >=65 years | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 184
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 203
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 203

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 4 in P2Y12 Reaction Units During Period 1
Description: The mean change in the P2Y12 reaction unit value assessed from baseline to the end of the 4-week maintenance dose treatment period, after switching from clopidogrel maintenance dose to prasugrel maintenance dose was analyzed with a paired t-test model. Mean changes (including standard deviations) are presented.
Time Frame: Baseline up to Week 4 post-maintenance dose prasugrel treatment period
Population: The P2Y12 reaction unit change from baseline was assessed in patients with available data in the Safety Population.
Measure: Mean (Standard Deviation); unit: P2Y12 reaction unit
Arm/Group | Prasugrel
Number analyzed (Participants) | 200
P2Y12 reaction unit | -18.2 (48.1)

2. Primary Outcome: Number of Participants With Thrombolysis In Myocardial Infarction (TIMI) Major Bleeding Events During Period 2
Description: All safety events were assessed in the overall Safety Population, regardless of the study period. The incidence of major bleeding events (defined as non-coronary artery bypass grafting [CABG] thrombolysis in myocardial infarction (TIMI) major) after 28 maintenance dose treatment weeks (optional maximum 12-month P2Y12 inhibitor treatment after ACS participants underwent PCI) are reported. Non-CABG TIMI major bleeding was defined as any intracranial bleeding (excluding microhemorrhages less than 10 millimeter evident only on gradient-echo magnetic resonance imaging); clinically overt signs of hemorrhage associated with a drop in hemoglobin of greater than or equal to 5 g/dL; and fatal bleeding (bleeding that directly results in death within 7 days)
Time Frame: End of Week 4 up to Week 28 post-maintenance dose prasugrel treatment period
Population: Number of participants with major bleeding events was assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prasugrel
Number analyzed (Participants) | 203
Participants | 4

3. Secondary Outcome: Number of Participants With High On-Treatment Platelet Reactivity (HTPR) During Period 1
Description: High On-Treatment Platelet Reactivity (HTPR) was defined as PRU >235.
Time Frame: Baseline up to Week 4 post-maintenance dose prasugrel treatment period
Population: High On-Treatment Platelet Reactivity was assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prasugrel
Number analyzed (Participants) | 203
Participants
  Baseline | 23
  Week 4 | 6

4. Secondary Outcome: Mean Percentage Change From Baseline to Week 4 in Platelet Inhibition During Period 1
Description: The mean percentage change in platelet inhibition at the end of the 4-week maintenance dose prasugrel treatment period, after switching from clopidogrel maintenance dose to prasugrel maintenance dose is reported.
Time Frame: Baseline up to Week 4 post-maintenance dose prasugrel treatment period
Population: Platelet inhibition was assessed in participants with available data in the Safety Population.
Measure: Mean (Standard Deviation); unit: percentage of platelet inhibition
Arm/Group | Prasugrel
Number analyzed (Participants) | 200
percentage of platelet inhibition | 7.2 (20.4)

5. Secondary Outcome: Number of Participants With Adverse Events of Special Interest During Period 1
Description: Adverse events of special interest were defined as major and minor bleeding events, clinically relevant bleeding events, and any major adverse cardiovascular events (MACE). Non-CABG TIMI major bleeding was defined as any intracranial bleeding (excluding microhemorrhages less than 10 millimeter evident only on gradient-echo magnetic resonance imaging); clinically overt signs of hemorrhage associated with a drop in hemoglobin of greater than or equal to 5 g/dL; and fatal bleeding (bleeding that directly results in death within 7 days). Non-CABG TIMI minor bleeding was defined as clinically overt (including imaging), resulting in hemoglobin drop of 3 to less than 5 g/dL.
Time Frame: Baseline up to Week 4 post-maintenance dose prasugrel treatment period
Population: Adverse events of special interest were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prasugrel
Number analyzed (Participants) | 203
Participants
  Any major bleeding adverse events (AE) | 0
  Any minor bleeding AE | 1
  Any clinically relevant bleeding AE | 2
  Any MACE, Cardiovascular death | 0
  Any MACE, Non-fatal myocardial infarction | 0
  Any MACE, Non-fatal stroke | 0
  Any MACE, Stent thrombosis | 0
  Any MACE, Revascularization | 0

6. Secondary Outcome: Number of Participants With Adverse Events of Special Interest During Period 2
Description: All safety events were assessed in the overall Safety Population, regardless of the study period. Adverse events of special interest were defined as major and minor bleeding events, clinically relevant bleeding events, and any major adverse cardiovascular events (MACE). Non-CABG TIMI major bleeding was defined as any intracranial bleeding (excluding microhemorrhages less than 10 millimeter evident only on gradient-echo magnetic resonance imaging); clinically overt signs of hemorrhage associated with a drop in hemoglobin of greater than or equal to 5 g/dL; and fatal bleeding (bleeding that directly results in death within 7 days). Non-CABG TIMI minor bleeding was defined as clinically overt (including imaging), resulting in hemoglobin drop of 3 to less than 5 g/dL.
Time Frame: End of Week 4 up to Week 28 post-maintenance dose prasugrel treatment period
Population: Adverse events of special interest were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Prasugrel
Number analyzed (Participants) | 203
Participants
  Any major bleeding AE | 4
  Any minor bleeding AE | 12
  Any clinically relevant bleeding AE | 4
  Any MACE, Cardiovascular death | 0
  Any MACE, Non-fatal myocardial infarction | 2
  Any MACE, Non-fatal stroke | 0
  Any MACE, Stent thrombosis | 0
  Any MACE, Revascularization | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the date of informed consent, and all adverse events which occurred after the first study medication intake and within 14 days after the treatment stop date was considered treatment emergent adverse events (TEAEs).
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding), symptom or disease, temporally associated with the use of a medicinal product, regardless of its nature, intensity, seriousness, or presumed relationship (causality) to the product or experimental procedure used.
Arm/Group | Prasugrel
All-Cause Mortality (participants affected / at risk) | 1/203
Serious Adverse Events (participants affected / at risk) | 28/203
Other Adverse Events (participants affected / at risk) | 125/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prasugrel (N=203)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Angina pectoris (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Hepatitis acute (Hepatobiliary disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Diverticulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Tonic convulsion (Nervous system disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic mass (Hepatobiliary disorders) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prasugrel (N=203)
Abdominal pain upper (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Dental caries (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Anal haemorrhage (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 2
Upper gastrointestional haemorrhage (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1
Gingival discomfort (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1
Oral disorder (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Tooth pulp haemorrhage (Gastrointestinal disorders) | 1
Angina pectoris (Cardiac disorders) | 7
Acute myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Chest pain (General disorders) | 6
Chest discomfort (General disorders) | 5
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Conjunctivitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Body tinea (Infections and infestations) | 1
Dermatophytosis of nail (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 4
Overdose (Injury, poisoning and procedural complications) | 3
Tendon injury (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Liver function test abnormal (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Weight increased (Investigations) | 1
Dizziness (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 3
Poor quality sleep (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Cerebral haemorrhage (Nervous system disorders) | 1
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Tonic convulsion (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 7
Dermatitis (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Haematuria (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 2
Nocturia (Renal and urinary disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Calculus bladder (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephritis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Thrombocytosis (Blood and lymphatic system disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Hepatitis (Hepatobiliary disorders) | 2
Hepatitis acute (Hepatobiliary disorders) | 2
Hepatic mass (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Vision blurred (Eye disorders) | 2
Ocular discomfort (Eye disorders) | 1
Breast tenderness (Reproductive system and breast disorders) | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Tooth extraction (Surgical and medical procedures) | 2
Stent placement (Surgical and medical procedures) | 1
Haematoma (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hypersensitivity (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT03672097/Prot_SAP_000.pdf